CLINICAL TRIAL: NCT06488794
Title: Inhaled Colistin to Prevent Pediatric Ventilator-associated Pneumonia: A Double Blind Multicenter Randomized Controlled Trial Protocol
Brief Title: Inhaled Colistin to Prevent Pediatric Ventilator-associated Pneumonia
Acronym: ColiPed
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Farah Thabet, PROFESSOR IN PEDIATRICS, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FThabet
Record Dates: First submitted 2024-06-15; First posted 2024-07-05 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Ventilator Associated Pneumonia
Keywords: colistin; mechanical ventilation; pneumonia; nebulization; prevention; pediatrics
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia | interventions — colistinmethanesulfonic acid; Colistin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- colistin group (Active Comparator): Colistin group:
  In the Nebulized colistimethate sodium (CMS) group, 100 000 IU/kg of CMS (equivalent to 0.96 mg/kg of colistin base), (maximum 750000 IU) will be nebulized daily, divided into two doses. The lyophilisate of CMS will be reconstituted as follows: 1 million of IU is reconstituted in 3 mL of sterile 0.9% saline. The adequate volume is then withdrawn and administered immediately to mechanically ventilated patients via a nebulizer until the nebulized solution container becomes empty.
  The nebulization is administered from day 3 of invasive mechanical ventilation, twice daily for a maximum of 7 days or until extubation (whichever occurres first).
  *12500 International Units of colistimethate sodium = 1 mg colistimethate sodium = 0.4 mg of colistin base.
  Interventions: Drug: colistimethate sodium
- Control group (Placebo Comparator): Nebulization of 3 ml of 0.9% saline twice a day for a maximum of 7 days from day 3 of invasive mechanical ventilation will be administered via a nebulizer until the nebulized solution container becomes empty.
  Interventions: Drug: 0.9% Saline

INTERVENTIONS:
Drug: colistimethate sodium — 100 000 IU/kg of colistimethate sodium (equivalent to 0.96 mg/kg of colistin base) ,maximum 750000 IU, will be nebulized daily, divided into two doses for a maximum of 7 days for eligible ventilated children starting from day 3 of mechanical ventilation.
  Other Names: Colistin
  Arms: colistin group
Drug: 0.9% Saline — Nebulization of 3 ml of 0.9% saline twice a day for a maximum of 7 days from day 3 of invasive mechanical ventilation for eligibile ventilated children
  Other Names: normal saline
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if nebulized colistimethate sodium can prevent pneumonia in ventilated children. The main question it aims to answer is:

• Does nebulized colistimethate sodium lower the number of times participants develop ventilation associated pneumonia? Researchers will compare nebulized colistimethate sodium to a placebo (a look-alike substance that contains no drug) to see if nebulized colistin works to prevent ventilation associated pneumonia in children.

Participants will:

* Take nebulized colistimethate sodium or a placebo twice a day for a maximum of 7 days.
* Will be followed to check for pneumonia occurrence while they are on mechanical ventilation.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the benefit of a 3 to 7 day course of inhaled colistimethate sodium among children undergoing invasive mechanical ventilation for more than 2 days on the occurrence of ventilator-associated pneumonia.

A double-blind, multicenter randomized controlled trial will be conducted. Patients on mechanical ventilation for more than 2 days will be randomized to receive inhaled colistin twice daily for 3 days or inhaled placebo (0.9% Sodium Chloride). Primary outcome will be the occurrence of ventilator-associated pneumonia from randomization to day 28.

ELIGIBILITY:
Inclusion Criteria:

* Children older than 1 month and younger than 14 years
* Patients on invasive mechanical ventilation for more than 48 hours
* Informed parental consent

Exclusion Criteria:

* Suspected or confirmed VAP on the day of inclusion
* Indication for systemic colistin therapy before or at enrolment in the study
* Plan for extubation within the next 24H
* Known allergy to colistin
* No parental consent
* Tracheostomy
* Appearance of allergic clinical manifestations in the days of colistin nebulization
* Appearance of undesirable clinical or biological manifestations presumed attributable to nebulization with colistin

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Ventilation Associated Pneumonia | From randomization to 28 days post-randomization
  Primary outcome will be the incidence of a first episode of ventilation associated pneumonia from randomization to day 28. Incidence will be calculated as the ratio of the number of patients experiencing a first VAP episode divided by the number of randomized patients

SECONDARY OUTCOMES:
Incidence of Ventilation Associated Tracheobronchitis | From randomization to 28 days post-randomization
  Incidence of first episode of ventilation associated tracheobronchitis (VAT) from randomization to day 28.
Incidence of a first episode of VAP and VAT in the subgroup of patients with tracheobronchial bacterial colonization at randomization | From randomization to 28 days post-randomization
  This secondary outcome measures the incidence of the first episode of ventilator-associated pneumonia (VAP) and ventilator-associated tracheobronchitis (VAT) within the first 28 days post-randomization in patients who had tracheobronchial bacterial colonization at the time of randomization. The 28-day period is selected to capture early occurrences of these infections and to evaluate the effectiveness of preemptive colistin nebulization in this high-risk subgroup.
Number of days spent on mechanical ventilation from randomization to day 28 | From randomization to 28 days post-randomization
  This secondary outcome measures the total number of days a patient remains on mechanical ventilation within the first 28 days following randomization. The 28-day period is chosen to assess the impact of preemptive colistin nebulization on reducing the duration of mechanical ventilation during the critical initial phase of ICU treatment.
Number of days without systemic antibiotics from randomization to day 28 | From randomization to 28 days post-randomization
  This secondary outcome measures the number of days without systemic antibiotic use within the first 28 days after randomization. The 28-day period is chosen to assess the impact of preemptive colistin nebulization on reducing the requirement for systemic antibiotics during the initial critical period of ICU treatment
ICU stay | From randomization to ICU discharge, up to 60 days
  Number of days spent in the ICU after randomization. This secondary outcome measures the length of stay in the ICU, defined as the number of days from randomization to ICU discharge. The time frame is chosen to comprehensively assess the duration of ICU treatment, which may be affected by the incidence of ventilator-associated pneumonia (VAP) and the impact of preemptive colistin nebulization on patient recovery
Incidence of antibiotic-resistant bacteria | From randomization to ICU discharge
  This secondary outcome measures the incidence of antibiotic-resistant bacteria isolated from routine clinical and hygiene samples collected from the date of randomization until ICU discharge. The time frame is chosen to monitor the development and prevalence of antibiotic-resistant bacteria throughout the entire ICU stay, providing insights into the impact of preemptive colistin nebulization on bacterial resistance patterns.
ICU day-28 mortality | 28 days from ICU admission
  This secondary outcome measures the mortality rate within 28 days of ICU admission. The time frame of 28 days is selected to assess early mortality outcomes related to ventilator-associated pneumonia and to evaluate the potential impact of preemptive colistin nebulization on patient survival during the initial critical period.

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: As soon as the manuscript is published
Access Criteria: request will be sent o the principal investigator by email, and will be shared if the reasons for request are academic or for planing similar study

REFERENCES:
- [Background] Zhu Y, Monsel A, Roberts JA, Pontikis K, Mimoz O, Rello J, Qu J, Rouby JJ; European Investigator Network for Nebulized Antibiotics in Ventilator-Associated Pneumonia (ENAVAP). Nebulized Colistin in Ventilator-Associated Pneumonia and Tracheobronchitis: Historical Background, Pharmacokinetics and Perspectives. Microorganisms. 2021 May 27;9(6):1154. doi: 10.3390/microorganisms9061154. PMID 34072189
- [Background] Jang JY, Kwon HY, Choi EH, Lee WY, Shim H, Bae KS. Efficacy and toxicity of high-dose nebulized colistin for critically ill surgical patients with ventilator-associated pneumonia caused by multidrug-resistant Acinetobacter baumannii. J Crit Care. 2017 Aug;40:251-256. doi: 10.1016/j.jcrc.2017.04.004. Epub 2017 Apr 7. PMID 28458172
- [Background] Karvouniaris M, Makris D, Zygoulis P, Triantaris A, Xitsas S, Mantzarlis K, Petinaki E, Zakynthinos E. Nebulised colistin for ventilator-associated pneumonia prevention. Eur Respir J. 2015 Dec;46(6):1732-9. doi: 10.1183/13993003.02235-2014. Epub 2015 Sep 24. PMID 26405294
- [Background] Povoa FCC, Cardinal-Fernandez P, Maia IS, Reboredo MM, Pinheiro BV. Effect of antibiotics administered via the respiratory tract in the prevention of ventilator-associated pneumonia: A systematic review and meta-analysis. J Crit Care. 2018 Feb;43:240-245. doi: 10.1016/j.jcrc.2017.09.019. Epub 2017 Sep 18. PMID 28942198